CLINICAL TRIAL: NCT02508272
Title: Transcriptomic Profiling in Severely Injured Patients
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Stv26/2007
Record Dates: First submitted 2015-07-20; First posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Trauma; Inflammation; Sepsis
Keywords: Transcriptome profiling
MeSH Terms: conditions — Wounds and Injuries; Inflammation; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — total RNA. Serum, Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trauma patients: age ≥18 y ISS ≥ 17 points admission < 6 h.

SUMMARY:
Discovery of differences in the host response in patients with systemic inflammation and sepsis, and identification of novel, specific markers by using a longitudinal clinico-transcriptomic approach.

DETAILED DESCRIPTION:
The aim of this study is to link defined clinical phenotypes with data on RNA obtained from blood samples by high throughput technologies. Genetic and molecular characteristics of the immune system after severe trauma will be crosslinked to clinical aspects of posttraumatic organ failure, with the goal of identifying typical molecular "fingerprints". Patients with and without sepsis or organ failure will be compared with the goal to develop a diagnostic test designed to predict the clinical course following severe trauma. Criteria for study enrollment includes patient age ≥18 y, an Injury Severity Score (ISS) ≥ 17 points, and time from injury to admission < 6 h. Whole blood from trauma patients will be collected within the first 6 h after trauma (day 0) and on days 1, 2, 3, 5, 7, 10, 14, and 21.

ELIGIBILITY:
Inclusion Criteria:

* patient age ≥18 y
* Injury Severity Score (ISS) ≥ 17 points
* time from injury to admission < 6 h.

Exclusion Criteria:

Moribund Patients with:

* PH < 7,1 or
* Lactate > 15 mmol/l or
* Base deficit > 15 mEq/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trauma patients with systemic inflammation due to multiple injuries (Polytrauma: ISS ≥ 17 points)
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2009-12; Primary Completion 2012-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Systemic Inflammation and Sepsis | 21 days after trauma

SECONDARY OUTCOMES:
Mortality | 28 days after Trauma
Nosocomial infections | 21 days after trauma
SOFA score | 21 days after trauma
Systemic inflammation score | 21 days after trauma
Hospital length of stay | 28 days after trauma
ICU length of stay | 28 days after trauma

CONTACTS AND LOCATIONS:
Overall Officials: Guido A Wanner, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Division of Trauma Surgery, Zurich, Switzerland